CLINICAL TRIAL: NCT05585086
Title: Determination of the Effect of Peppermint Oil Inhalation on Postoperative Nausea, Vomiting and Comfort
Brief Title: Effect of Peppermint Oil Inhalation on Postoperative Nausea, Vomiting and Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gümüşhane Universıty (Other)
Collaborators: Kırklareli University (Other)
Responsible Party: Principal Investigator, Nursen Kulakac, Principal Investigator, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GumushaneU2
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Inhalation; Oil
Keywords: patient; nausea; Vomiting; mentha piperita; postoperative
MeSH Terms: conditions — Respiratory Aspiration; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Peppermint oil will be applied by diluting 1/10 in wheat oil so that it does not cause skin irritation.
  Interventions: Other: Peppermint Oil Inhalation
- Control (No Intervention): Patients who underwent surgery will be monitored for the severity of nausea and vomiting after surgery. Follow-ups are 0-2, 2-6, 6-12, 12-24 and 24-48 postoperatively. hours and will be recorded without any application or intervention by the researcher.

INTERVENTIONS:
Other: Peppermint Oil Inhalation — Peppermint oil will be given by diluting 1/10 in wheat oil so that it does not cause skin irritation. Application; by inhalation method, 2 cc lavender essential oil + 100 cc water (2%) will be in the form of two drops for 20 minutes. Since the effectiveness of essential oils decreases over time and the desired dose cannot be applied at the same time; Peppermint oil will be applied to the individual for a total of 5 times every 30 minutes.
  Arms: Experimental

SUMMARY:
Nausea and vomitting related to drugs and anesthetic methods are among the important postoperative problems. Nausea and vomitting causing illlness feeling of patient are frequent after surgical interventions, cause increased dissatisfaction of the patient and prolonged discharge period. In this study it was aimed to evaluate the effect of peppermint oil inhalation on postoperative nausea and vomitting.

Purpose and Type of Research The randomized controlled study will be performed on patients undergoing laparoscopic cholecystectomy, which is the most commonly performed surgical procedure, in a general surgery clinic of a training and research hospital.

DETAILED DESCRIPTION:
Nausea and vomitting related to drugs and anesthetic methods are among the important postoperative problems. Nausea and vomitting causing illlness feeling of patient are frequent after surgical interventions, cause increased dissatisfaction of the patient and prolonged discharge period. In this study it was aimed to evaluate the effect of peppermint oil inhalation on postoperative nausea and vomitting. Purpose and Type of Research The randomized controlled study will be performed on patients undergoing laparoscopic cholecystectomy, which is the most commonly performed surgical procedure, in a general surgery clinic of a training and research hospital.

Location of the research This research will be carried out in a 24-bed general surgery clinic of a 250-bed training and research hospital located in western Turkey. In the Surgery Service, nurses work in three shifts, 08:00-16:00, 16:00-24:00 and 24:00-08:00, while the responsible nurse works between 08:00-17:00. In the surgical service, there are a total of 24 patient rooms, all of which are single beds. Clinical routines in the surgery clinic include pharmacological methods and there is no use of complementary therapy methods.

Population and Sample of the Research 60 patients are planned to be included in the study. In the creation of randomization; Experiment and control group will be assigned by computer method. In this way, experimental applications will be continued until the number of patients in both groups is completed. During the trial period, patients who wish to withdraw or need to be excluded from the trial will be excluded.

Research Hypotheses H0. Peppermint oil inhalation has no effect on post-operative nausea. H1. Peppermint oil inhalation has an effect on post-operative nausea. H0. Peppermint oil inhalation has no effect on postoperative comfort. H0. Peppermint oil inhalation has an effect on postoperative comfort.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old, 65 years old and under,
* having colonoscopy,
* not having the risk of heart failure and cardiogenic shock (class III and IV),
* not having a history of asthma, eczema and allergies to flowers and plants,
* no peppermint oil allergy,
* no communicative / severe hearing or speech impairment,
* no use of antidepressant, antihistamine, diuretic, hypnotic, benzodiazepine and narcotic derivatives
* ASA score of 1 or 2
* Individuals willing to participate will be included in the study.

Exclusion Criteria:

• Individuals who do not meet the inclusion criteria will not be included in the

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Nause | 7 day
  post-operative nausea rate

IPD SHARING:
Plan to Share IPD: No